CLINICAL TRIAL: NCT04341467
Title: Amisulpride Versus Olanzapine Treatment for Behavioral and Psychological Symptoms in Patients With Dementia of the Alzheimer Type:A Randomized, Open-label, Prospective Study
Brief Title: Amisulpride Treatment for BPSD in AD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMI-2019-BPSD
Record Dates: First submitted 2019-12-27; First posted 2020-04-10 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: BPSD; Amisulpride; Olanzapine; Dementia of the Alzheimer Type
MeSH Terms: interventions — Amisulpride; Olanzapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amisulpride group (Experimental): The initial dose of amisulpride group is 50mg/d, and the maximum dose is 800mg/d.
  Interventions: Drug: Amisulpride
- Olanzapine group (Active Comparator): The initial dose of olanzapine is 2.5 mg/d, and the maximum dose is 20 mg/d.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Amisulpride — The initial dose of amisulpride group is 50mg/d, and the maximum dose is 800mg/d.
  Other Names: Solian
  Arms: Amisulpride group
Drug: Olanzapine — The initial dose of olanzapine is 2.5 mg/d, and the maximum dose is 20 mg/d.
  Other Names: Oulanning
  Arms: Olanzapine group

SUMMARY:
Currently, olanzapine is the most widely used and studied drug for the treatment of behavioral and psychological symptoms in patients with Alzheimer's disease, but there are significant side effects. Amisulpride is a new antipsychotic that not only controls mental symptoms but also improves cognitive function. Therefore, the aim of this study was to evaluate the effectiveness and tolerability of both amisulpride and Olanzapine for treating the behavioral and psychological symptoms of dementia in patients with dementia of the Alzheimer type.

DETAILED DESCRIPTION:
This study was a randomized, open-label, prospective clinical study in which patients were randomized to receive amisulpride and olanzapine for 8 weeks. Drug efficacy and safety assessments were assessed at baseline, 2 weekends, 4 weekends, and 8 weekends.

ELIGIBILITY:
Inclusion Criteria:

1. It conforms to the diagnostic standard of Alzheimer's disease in International Classification of Diseases 10th Revision (ICD-10)
2. a total score of MMSE<24
3. The patients had active behavioral symptoms with a minimum score of 20 on the 12-point Neuropsychiatric Inventory (NPI)
4. Participant or guardian has to sign informed consent. The patients' guardians will sign the informed consent on behalf of the participants when the capacity of participants to consent is compromised

Exclusion Criteria:

1. People with vascular dementia, frontotemporal dementia, dementia with Lewy bodies or other neurocognitive disorders;
2. Patients with severe brain organic diseases or brain trauma;
3. Physical illnesses associated with severe respiratory, circulatory, immune, and endocrine systems;
4. History of other mental disorders;
5. Those who are allergic to amisulpride or olanzapine;
6. Patients who are contraindicated with amisulpride and olanzapine: pheochromocytoma, prolactin-dependent tumors and narrow-angle glaucoma;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes of neuropsychiatric inventory（NPI）scores | baseline, Week 2,4, and 8
  The change from baseline neuropsychiatric inventory (NPI) items at week 2,4,and 8. Assess the frequency and severity of psychiatric symptoms, including delusions, hallucinations, aggression attacks, depression, anxiety, elevated emotions, indifferent emotions, de-inhibition, agitation, abnormal behaviors, sleep / night behaviors, appetite / eating disorders,the maximum scores is 144.The higher score are considered the psychiatric symptoms more serious.

SECONDARY OUTCOMES:
Changes of Clinical global impression-Severity of Illness (CGI-SI) score | baseline, Week 2,4, and 8
  The change from baseline Clinical global impression-Severity of Illness (CGI-SI) score.
  The highest score is 7 points. A higher score indicates a more serious disease or a tendency to worsen The change from baseline Clinical global impression-Severity of Illness (CGI-SI) score.
  The highest score is 7 points. A higher score indicates a more serious disease or a tendency to worsen
Changes of Clinical global impression- global improvement (CGI-GI) | baseline, Week 2,4, and 8
  The change from baseline Clinical global impression- global improvement (CGI-GI) items at week 2,4,and 8.
  The highest score is 7 points. A higher score indicates a more serious disease or a tendency to worsen
Changes of Mini-Mental State Examination(MMSE) scores. | baseline, Week 2,4, and 8
  The change from baseline Mini-Mental State Examination(MMSE) items at week 2,4,and 8.The content includes time orientation, location orientation, immediate memory of language, attention and calculation, short-term memory, physical naming, language repeating, reading comprehension, speech expression and graphic description. 0 to 30 points, the lower the score, the more severe the cognitive impairment.
Changes of Caregiver Burden Inventory (CBI) scores | baseline, Week 2,4, and 8
  The change from baseline Caregiver Burden Inventory (CBI) items at week 2,4,and 8.The questionnaire contains 5 dimensions: time-dependent burden, development-restricted burden, physical burden, social burden, and emotional burden. The total score is 96 points. The higher the score, the heavier the burden.
Treatment Emergent Symptom Scale (TESS) | Week 2,4, and 8
  The scale collection includes 33 items of consciousness disorder, constipation, tremor, etc., to assess the adverse drug reactions and their severity.This table is used to evaluate 33 items of common consciousness disorder, constipation, tremor, etc. based on the adverse drug reactions. Each item is scored according to the severity of the adverse drug reactions. This scale does not need to be evaluated at baseline.
Rating scale for extrapyramidal side effects (RSESE) | baseline, Week 2,4, and 8
  Assessment of extrapyramidal reactions and their severity at various time points.Assess the severity of 9 aspects of gait, falling arms, shaking shoulders, elbow rigidity, fixed posture or wrist rigidity, leg swings, head and neck movements, tapping between eyebrows, drooling，The total score is 36 points. The higher the score, the more severe extrapyramidal side effects.
Abnormal Involuntary Movement Scale (AIMS) | baseline, Week 2,4, and 8
  Assesses whether patients have involuntary movements and their severity in the face, limbs, and trunk at various time points.Assess facial movements, body movements, and trunk movements for involuntary movements and severity. A total score of 2 or more is masculine gender.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China